CLINICAL TRIAL: NCT06275425
Title: Comparison of the Coughing Frequency of Remimazolam Total Intravenous Anesthesia Versus Inhalational Anesthesia : a Single-blinded Randomized Controlled Trial
Brief Title: Comparison of the Coughing Frequency of Remimazolam Total Intravenous Anesthesia Versus Inhalational Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2023-0429
Record Dates: First submitted 2023-12-12; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Thyroid Neoplasm; Cough
MeSH Terms: conditions — Thyroid Neoplasms; Cough | interventions — Anesthesia, Inhalation; Sevoflurane

STUDY DESIGN:
Intervention Model Description: a single-blinded randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): General anesthesia is maintained with intravenous administration of Byfavo.
  Interventions: Drug: Total intravenous anesthesia with Byfavo
- Control (Active Comparator)
  Interventions: Drug: Inhalation anesthesia with Sevoflurane

INTERVENTIONS:
Drug: Total intravenous anesthesia with Byfavo — General anesthesia is maintained with intravenous continuous administration of Byfavo.
  Arms: Intervention
Drug: Inhalation anesthesia with Sevoflurane — General anesthesia is maintained with Sevoflurane.
  Arms: Control

SUMMARY:
This study is a randomized controlled trial. Adult patients undergoing thyroidectomy under general anesthesia at Severance Hospital and Yonsei Cancer Center are included in tis study. For intervention group, patients receive anesthesia with total intravenous remimazolam, while for control group, patients receive anesthesia with inhalation anesthetic.

The primary end point of the study is to determine whether coughing during endotracheal tube extubation is less when anesthesia is maintained with intravenous remimazolam compared to inhalation anesthetics. The secondary end points are cough score (graded into 4 levels), frequency of reoperation due to postoperative bleeding, These include the frequency of hypertension during the extubation process and whether additional painkillers are used in the recovery room.

ELIGIBILITY:
Inclusion Criteria:

Adult patients aged 19 years or older undergoing thyroidectomy under general anesthesia at Severance Hospital Cancer Center.

Exclusion Criteria:

* Patients with American society of anesthesiologists physical status classification IV or higher.
* Patients who are hypersensitive to remimazolam or inhalational anesthetic.
* Patients with structural abnormalities in the upper airway or respiratory diseases.
* Patients with a history of upper respiratory tract infection within the past 2 weeks.
* Current smoker
* Pregnant
* Patients who have difficulty reading and understanding the informed consent form

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-06-25 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients not coughing during postoperative extubation | Until discharge (3days on average)
  Proportion of patients not coughing during postoperative extubation

SECONDARY OUTCOMES:
Cough score | Until discharge (3days on average)
  Cough score (4 scale score: 1- no cough, 2: cough once, 3: cough lating less than 5 seconds, 4: cough lating longer than 5 seconds.)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Joung No, Principal Investigator — Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, College of Medicine, Yonsei University, Seoul
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, College of Medicine, Yonsei University,, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No